CLINICAL TRIAL: NCT05424562
Title: Capturing Canadian Real-World Data for AML Chemotherapy Ineligible Patients on Venetoclax (LIVEN)
Brief Title: A Study to Assess Change in Disease State in Adult Participants With Acute Myeloid Leukemia (AML) Ineligible for Intensive Chemotherapy Receiving Oral Venetoclax Tablets in Canada
Acronym: LIVEN
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-363
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Venclexta; Venclyxto; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants treated with Venetoclax in accordance with approved local label.

SUMMARY:
Acute Myeloid Leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well venetoclax works to treat AML in adult participants who are ineligible for intensive induction chemotherapy in Canada.

Venetoclax is a drug approved to treat Acute Myeloid Leukemia (AML). All study participants will receive Venetoclax as prescribed by their study doctor in accordance with approved local label. Adult participants with a new diagnosis of AML who are ineligible for intensive induction chemotherapy will be enrolled. Around 200 participants will be enrolled in the study in approximately 15-20 sites in Canada.

Participants will receive venetoclax tablets to be taken by mouth daily according to the approved local label. The duration of the study is approximately 36 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute Myeloid Leukemia (AML).
* Ineligible for intensive chemotherapy, determined by the physician's assessment of age, Eastern Cooperative Oncology Group Performance Status (ECOG-PS), comorbidities, regional guidelines, and institutional practice.
* Participant for whom the physician has decided to initiate venetoclax treatment in accordance with the local label. The decision to treat with venetoclax is made by the physician prior to any decision to approach the participant to participate in this study.

Exclusion Criteria:

- Participation in an interventional clinical trial within 30 days prior to venetoclax treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with acute myeloid leukemia (AML) treated with venetoclax per approved local label in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 36 Months
  OS as defined by number of days from start of treatment to the completion of treatment or death from any cause.

SECONDARY OUTCOMES:
Change in Composite Complete Remission Rate | Up to 36 Months
  Composite Complete Remission Rate is defined as complete remission (CR) plus complete remission with incomplete hematologic recovery (CRi) as described by the modified International Working Group (IWG) criteria.
Event-Free Survival (EFS) | Up to 36 Months
  EFS as defined by number of days from start of treatment to the date of progressive disease, relapse from CR or CRi, treatment failure or death from any cause.
Percentage of Participants with Presence Transfusion Independence | Up to 36 Months
  Transfusion Independence is defined as at least 8 and/or 16 consecutive weeks without an Red Blood Cell (RBC) or platelet transfusion during the treatment period.
Number of Participants with Transfusions | Up to 36 Months
  Number of Participants with transfusions (red blood cells and platelets).
Number of Participants with Change in Venetoclax Dose | Up to 36 Months
  Number of participants with change in venetoclax dose.
Number of Participants with Change in Other Medications | Up to 36 Months
  Number of participants with change in other medications.
Venetoclax Administration Setting | Up to 36 Months
  Venetoclax administration setting (in-patient vs. out-patient vs. at home).
Number of Hospital Admission | Up to 36 Months
  Number of hospital admission.
Number of Participants with Change in use of Antiinfectives | Up to 36 Months
  Number of participants with change in use of antiinfectives.
Number of Participants with Change in Tumor Lysis Syndrome (TLS) Risk | Up to 36 Months
  Number of participants with change in TLS risk.
Occurrence of any Adverse Events | Up to 36 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with their treatment as graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (20):
- Canada (20):
  - Tom Baker Cancer Centre /ID# 248113, Calgary, Alberta
  - University of Alberta Hospital /ID# 251531, Edmonton, Alberta
  - BC Cancer - Surrey /ID# 257515, Surrey, British Columbia
  - Vancouver General Hospital /ID# 245438, Vancouver, British Columbia
  - BC Cancer - Victoria /ID# 257339, Victoria, British Columbia
  - CancerCare Manitoba /ID# 246414, Winnipeg, Manitoba
  - The Moncton Hospital /ID# 247277, Moncton, New Brunswick
  - Eastern Regional Health Authority /ID# 250241, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 246514, Halifax, Nova Scotia
  - Juravinski Cancer Centre /ID# 247183, Hamilton, Ontario
  - Kingston Health Sciences Centre /ID# 253439, Kingston, Ontario
  - London Health Sciences Center- University Hospital /ID# 248027, London, Ontario
  - Lakeridge Health - Oshawa /ID# 246412, Oshawa, Ontario
  - Thunder Bay Regional Research Institute /ID# 249163, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre /ID# 251966, Toronto, Ontario
  - University Health Network_Princess Margaret Cancer Centre /ID# 249607, Toronto, Ontario
  - Disc_Royal Victoria Hospital / McGill University Health Centre /ID# 249704, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 248915, Sherbrooke, Quebec
  - Allan Blair Cancer Centre /ID# 247663, Regina, Saskatchewan
  - Saskatoon Cancer Centre /ID# 247181, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.rxabbvie.com/